CLINICAL TRIAL: NCT05741229
Title: The Effect Of Nebulizied Nitroglycerin As An Adjuvant Drug In Management Of Persistent Pulmonary Hypertension Of Newborns
Brief Title: The Effect Of Nebulizied Nitroglycerin As An Adjuvant Therapy For Persistent Pulmonary Hypertension Of Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Primary Investigator and Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201737
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn; Echocardiography; Respiratory Disease
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome; Respiration Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (nebulized nitroglycerine) (Active Comparator): Patients with persistent pulmonary hypertension (PPHN) and will receive nebulized nitroglycerine as an adjuvant therapy for PPHN
  Interventions: Drug: Nebulized nitroglycerine as adjunctive therapy
- Group II (conentional treatment group) (Placebo Comparator): Patients with PPHN and will be treated with conventional regimen for PPHN
  Interventions: Drug: conventional therapy for PPHN

INTERVENTIONS:
Drug: Nebulized nitroglycerine as adjunctive therapy — Patients with PPHN will have nebulized nitroglycerine as adjunctive therapy
  Arms: Group I (nebulized nitroglycerine)
Drug: conventional therapy for PPHN — patients will receive sildenafil which is used routinely in management of PPHN in our unit, in addition to appropriate oxygenation and ventilation.
  Arms: Group II (conentional treatment group)

SUMMARY:
This aim of the study is to evaluate the effect of nebulized nitroglycerin on echocardiographic (biventricular function, pulmonary artery pressure, PDA and PFO shunting and tissue doppler imaging) and clinical parameters (Oxygen saturation index, heart rate, blood pressure, mean airway pressure, ventilation setting) in patients with PPHN.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≤72 hours' old, ≥37 weeks of gestation, ≥50% FiO2 need despite lung recruitment, abnormal oxygen saturation index or echocardiographic signs of PPHN will be enrolled in the trial.

Exclusion Criteria:

* • Diagnosis of PPHN discovered after more than 72 hours.

  * Failure of used medications and need to administrate milrinone

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Estimation of Pulmonary artery pressure (PAP) | first 7 days of life
  Systolic pulmonary artery pressure (SPAP) can be estimated by measuring the peak velocity of tricuspid valve regurgitation with the use of the modified Bernoulli's equation.
  * The estimation of SPAP by measuring TR is reliable and often equivalent to pressures measured in the catheter lab while using continuous wave Doppler. However, the accuracy depends on the quality of the acquired TR jet. An optimal quality TR jet shows a well demarcated envelope.
  * Right atrial pressure (RAP) is usually not measured, and a value of 3- 5 mmHg is generally assumed.
Right ventricular (RV) function in ml/kg/min | first 7 days of life
  • RV output and stroke distance in main pulmonary artery:
  * CSA (cm) (Cross sectional area of PV by long axis parasternal RV outflow view - 2D - immediately beneath pulmonary annulus - mid-systole - inner edge to inner edge) = π x (radius)2 ✓ VTI (cm) (Velocity Time Integral or Stroke Distance = Distance over which blood travels in once cardiac cycle → Long axis parasternal RV outflow view). 12. ✓ SV (ml/beat) (Stroke Volume = CSA x VTI).
  * Output (L/min.) COP = SV x HR.
Left ventricular (LV)function in ml/kg/min | first 7 days of life
  LV output and stroke distance in ascending aorta:
  * CSA (cm) (Cross sectional area of AV by long axis parasternal view - 2D - immediately beneath aortic annulus - mid- systole - inner edge to inner edge) = π x (radius)2. ✓ VTI (cm) (Velocity Time Integral or Stroke Distance = Distance over which blood travels in once cardiac cycle → Apical 5-chamber view).
  * SV (ml/beat) (Stroke Volume = CSA x VTI).
  * Output (L/min.) COP = SV x HR.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Ghazal, PhD, Study Chair — Alexandria University; Aly Mohamed Abdel-Mohsen, PhD, Study Director — Alexandria University; Moataz Shawky Rezk, MD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data is available for meta-analysis or any useful study upon reasonable request to authors
Supporting Information: Study Protocol
Time Frame: 6 years after termination of study
Access Criteria: available on reasonable request to researcher

REFERENCES:
- [Background] Bethou A. Utility of Nebulized Magnesium Sulfate Therapy for Persistent Pulmonary Hypertension of Newborn. Indian J Pediatr. 2021 Aug;88(8):749-750. doi: 10.1007/s12098-021-03851-0. Epub 2021 Jun 23. No abstract available. PMID 34164785
- [Derived] Farag MM, Ghazal HAE, Abdel-Mohsen AM, Rezk MA. Nebulized nitroglycerin as an adjuvant drug in management of persistent pulmonary hypertension of newborns: a randomized controlled trial. Eur J Pediatr. 2025 Sep 1;184(9):586. doi: 10.1007/s00431-025-06381-5. PMID 40888971
- See also: Idea about neubilized medications in PPHN — https://pubmed.ncbi.nlm.nih.gov/34164785/